CLINICAL TRIAL: NCT04203108
Title: ATG Used in Allogeneic Hematopoietic Stem Cell Transplantation From HLA-matched Sibling Donor as GVHD Prophylaxis
Brief Title: ATG in HLA-matched Sibling HSCT as GVHD Prophylaxis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Principal Investigator, Qifa Liu, Professor, Nanfang Hospital, Southern Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATG in HLA-matched HSCT-2019
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Hematopoietic Stem Cell Transplantation
Keywords: Hematopoietic Stem Cell Transplantation; antithymocyte globulin; graft-versus-host disease
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATG group (Experimental): ATG group refers to treatment with a protocol including low-dose ATG, CsA, short-term MTX and MMF as GVHD prophylaxis.
  Interventions: Drug: ATG; Drug: CsA; Drug: MTX; Drug: MMF
- non-ATG group (Active Comparator): Non-ATG group refers to treatment with a protocol including CsA, short-term MTX and MMF as GVHD prophylaxis.
  Interventions: Drug: CsA; Drug: MTX; Drug: MMF

INTERVENTIONS:
Drug: ATG — In ATG group, ATG will be intravenously infused via a central venous catheter in day -1 at a dose of 2.5mg/kg.
  Arms: ATG group
Drug: CsA — In both groups, CsA will be intravenously infused from day -9 and the dose was adjusted based on the concentration.
Drug: MTX — In both groups, MTX will be intravenously on days +1(15mg), +3(10mg) and +6(10mg).
Drug: MMF — In both groups, MMF will be administrated at a dose of 1.0g/d.

SUMMARY:
The protocols including ciclosporin A （CsA）+methotrexate (MTX) +mycophenolate Mofetil(MMF) have been widely used for graft-versus-host disease (GVHD) prophylaxis in allogeneic hematopoietic stem cell transplantation from HLA-matched sibling donor (MSD). Nevertheless, severe chronic graft-versus-host disease (cGVHD) remains an obstacle for MSD HSCT. A growing body of studies have suggested antithymocyte globulin (ATG) could reduce the incidence of cGVHD. This study is aim to evaluate the efficacy of a protocol that includes CsA, MTX, MMF and ATG in recipients of MSD HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. A patient age of 18-65 years
2. MSD transplant recipient
3. Subjects (or their legally acceptable representatives) must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

1. Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
2. Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 266 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
the incidence of cGVHD | 2 year posttransplantation
  cGVHD was graded as limited or extensive.

SECONDARY OUTCOMES:
overall survival | 2 year posttransplantation
disease-free survival | 2 year posttransplantation
the incidence of aGVHD | 100 days 1 year posttransplantation
  aGVHD was defined according to the 1994 Consensus Conference on Acute GVHD Grading and graded from I to IV.

CONTACTS AND LOCATIONS:
Overall Officials: Qifa Liu, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided